CLINICAL TRIAL: NCT02318654
Title: Comparing the Efficacy of Ice Pack Versus Topical EMLA for Pain Control in Laser Axillary Hair Removal: A Randomized Control Trial
Brief Title: Ice Versus EMLA for Pain in Laser Hair Removal
Status: Active, not recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Northwestern University (Other)
Responsible Party: Principal Investigator, Murad Alam, Professor in Dermatology, Otolaryngology-Head and Neck Surgery, and Surgery, Northwestern University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: STU106090
Record Dates: First submitted 2014-12-12; First posted 2014-12-17 (Estimated); Last update posted 2025-01-31 (Actual); Status verified 2025-01

CONDITIONS: Hair Removal
MeSH Terms: interventions — Lidocaine, Prilocaine Drug Combination

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Ice Pack (Active Comparator)
  Interventions: Other: Ice Pack
- Topical EMLA cream (Active Comparator)
  Interventions: Drug: Topical EMLA cream

INTERVENTIONS:
Other: Ice Pack — Subjects will have 600 grams of ice in clear plastic bag size 18 x 23 cm applied to the randomized axilla for 10 minutes. After 10 minutes, the ice pack will be removed and laser hair treatment will be performed.
  Arms: Ice Pack
Drug: Topical EMLA cream — Topical EMLA will be applied approximately 2 mm thick to the randomized axilla with a wooden tongue depressor wrapped with impermeable plastic occlusion dressing for 60 minutes. After 60 minutes, the drug will be removed with regular gauze and saline and laser hair treatment will be performed.
  Arms: Topical EMLA cream

SUMMARY:
The primary objective of this study is to compare the efficacy of ice pack to topical eutectic mixture of local anesthesia (EMLA) for pain control in diode 810 nm laser axillary hair removal.

This study is a pilot study designed to determine feasibility of these procedures.

ELIGIBILITY:
Inclusion Criteria

1. Subjects are Caucasian or Asian females.
2. Subjects are 18-65 years old.
3. Subjects have Fitzpatrick skin type I-III and coarse dark axillary hair.
4. Subjects are in good health.
5. Subjects can provide informed consent.
6. Subjects have the willingness and the ability to understand and communicate with the investigators.

Exclusion Criteria

1. Subjects who are allergic to lidocaine or prilocaine.
2. History of methemoglobinemia.
3. History of recurrent petechial or purpuric lesions.
4. Bleeding tendency or coagulopathy.
5. History of laser treatment in axilla.
6. History of keloid or hypertrophic scarring.
7. Pregnant or lactating or intends to become pregnant in the next 3 months.
8. Active skin disease or skin infection in the treatment area.
9. Subjects with known mental illness or other psychological conditions, such as psychotic disorders, mood disorders, anxiety disorders and cognitive disorders.
10. History of cold urticaria.
11. History of current injury or abnormal skin sensation.
12. Unable to understand the protocol or to give informed consent.
13. Any other condition that would, in the professional opinion of the investigator, potentially affect response or participation in the clinical clinical study, or would pose as an unacceptable risk to subject.

Ages: 18 Years to 65 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2014-12-30 (Actual); Primary Completion 2025-12 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Pain using the SF-MPQ immediately after treatment | immediately (at 0 min) after laser treatment
Pain using the SF-MPQ 5 minutes after treatment | 5 mins after laster treatment

CONTACTS AND LOCATIONS:
Overall Officials: Murad Alam, MD, Principal Investigator — Northwestern University
Locations (1):
- Northwestern University Feinberg School of Medicine, Department of Dermatology, Chicago, Illinois, United States